CLINICAL TRIAL: NCT06877663
Title: Impact of Virtual Reality on Anxiety Management During Elective Surgery
Brief Title: Virtual Reality on Anxiety Management During Elective Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Claudio Gambardella, Associate Professor, MD, PhD, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Virtual Reality
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Discomfort; Pain Intensity Assessment
Keywords: Anxiety; Virtual Reality; Preoperative management; Postoperative Pain
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This is a prospective, low-interventional randomized study on consecutive patients candidates for elective surgery. To investigate the effect of preoperative Virtual Reality (VR) entertainment on patient anxiety, patients will be randomized into two groups:
  * Group A: Patients who will receive entertainment videos via VR headset in the preoperative room before surgery.
  * Group B: Patients who will receive standard preoperative care and will serve as the control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and Outcome Assessor were all blinded to treatment allocation. Because the blinding of the operating surgeons was not feasible, they were not involved in the data collection and outcome assessment. Physicians in charge of patients' management were not involved in the operating room and were blinded to the device use. The data were collected and analyzed by physicians who were not involved in the patient's management during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Group (Experimental): Group A: Patients who will receive entertainment videos via VR headset in the preoperative room before surgery.
  Interventions: Device: Virtual Reality Device
- Control Group (No Intervention): Group B: Patients who will receive standard preoperative care and will serve as the control group.

INTERVENTIONS:
Device: Virtual Reality Device — Patients who will receive entertainment videos via VR headset in the preoperative room before surgery.
  Arms: Virtual Reality Group

SUMMARY:
The aim of this research is to assess and compare the effects of audiovisual content administered via specific Meta Quest 2 headsets on pre-surgical anxiety in patients undergoing elective surgical procedures and on procedure-related comfort.

DETAILED DESCRIPTION:
Preoperative anxiety is a very common condition in all individuals undergoing surgical procedures. On the day of the procedure, in fact, between 50% and 70% of patients experience anxiety, which usually peaks during anesthesia induction. The main concerns underlying pre-surgical anxiety include fear of surgical complications, worries about the duration of the procedure, the potential onset of subsequent disabilities, as well as concerns regarding general anesthesia and the associated loss of control. Additionally, a common fear is waking up and experiencing discomfort and pain during the procedure. More anxious patients are at greater risk of problems during anesthesia induction, difficulties in pain management, and a more challenging recovery. These frequent conditions highlight the need for interventions aimed at reducing preoperative anxiety.

Currently, the most common prevention/treatment for preoperative anxiety is a pharmacological approach. The pharmacological option includes sedatives and anxiolytic drugs, which, however, may cause adverse effects such as respiratory problems, drowsiness, interactions with anesthetic drugs, and prolonged recovery time. Therefore, non-pharmacological interventions are becoming increasingly common.

There are also other non-pharmacological approaches, although less widespread, including cognitive-behavioral therapy (the current gold-standard treatment for anxiety disorders), aromatherapy, and music therapy. Additionally, in pediatric surgery, audiovisual support has been tested as a means of reducing anxiety levels, particularly when focused on providing preoperative management information, administered 48 hours before the scheduled surgery. This practice has also been found to be more satisfactory than traditional play activities with toys.

Currently, several all-in-one virtual reality (VR) headsets are available on the market, capable of immersing an individual in an artificially constructed reality. Specifically, the Meta Quest 2 ™ headset (Meta®, Menlo Park, California, USA) explores VR on a standalone platform, with advanced privacy features to encrypt data and parental supervision tools to ensure appropriate content for all users. In the medical field, VR headsets have already been tested in rehabilitation, ophthalmology, and surgery as a therapeutic method for patients, as well as a fundamental tool for physician training.

The objective of this study is to evaluate the impact of VR on patients undergoing elective surgery in reducing preoperative anxiety and improving patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Age <70 years
* Indication for elective surgery

Exclusion Criteria:

* Diagnosis of Anxiety Disorder, Major Depression, Personality Disorder, Bipolar Syndrome
* Substance abuse
* Inability to complete the study protocol
* Patients for whom the surgical procedure was not performed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
STAI score | It will be administered at three different time points for both the control group (Group B) and the experimental Group A (screening, before surgery, and 48 hours after the operation) to quantify patient anxiety levels.
  Assessment of the difference in State-Trait Anxiety Inventory (STAI; range 20-80; a higher score indicates a higher level of anxiety) score between the two groups at baseline, preoperatively, and postoperatively

SECONDARY OUTCOMES:
VAS scale | It will be evaluated at 12-24-48 hours after surgery
  Perioperative pain will be evaluated using the Visual Analog Scale (VAS; range 0-10; a higher score indicates greater pain).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania Luigi Vanvitelli, Caserta, CE, Italy

IPD SHARING:
Plan to Share IPD: Undecided
We have to discuss it with the central Institution